CLINICAL TRIAL: NCT03984903
Title: Learning of Motor Control Exercises With Different Methods and Its Effects on Treatment Outcomes in Patients With Chronic Non-specific Low Back Pain: A Randomised Controlled Trial
Brief Title: Different Learning Methods of Motor Control Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Utku BERBEROĞLU, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-180060
Record Dates: First submitted 2019-05-30; First posted 2019-06-13 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Back Pain Without Radiation
Keywords: Back Pain without Radiation; Low Back Pain, Mechanical
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face Learning Group (Active Comparator)
  Interventions: Other: Face-to-face Learning of Exercises; Other: Manual Therapy; Other: Home Exercise Program
- Multimedia Learning Group (Experimental)
  Interventions: Other: Multimedia Learning of Exercises; Other: Manual Therapy; Other: Home Exercise Program

INTERVENTIONS:
Other: Multimedia Learning of Exercises — Patients learn exercise from multimedia content.
  Arms: Multimedia Learning Group
Other: Face-to-face Learning of Exercises — Physiotherapist teach exercises to patients
  Arms: Face-to-face Learning Group
Other: Manual Therapy — Myofascial Release Techniques and Joint Mobilizations to the Lumbal Area
Other: Home Exercise Program — Patients do at least 20 minutes motor control exercise in a day at home.

SUMMARY:
This study evaluates the effects of self-learning exercise from multimedia content on pain and disability in patients with low back pain.

DETAILED DESCRIPTION:
For see the full effect of exercise treatment, exercise adherence should be high. In patients with chronic non-specific low back pain, the complex nature of the core-stabilization exercises decrease the exercise adherence. Some novel studies show that multimedia learning can increase efficiancy of complex skill learning and can be better from classic face to face learning.

So this study evaluates the effects of self-learning exercise from multimedia content on pain and disability in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (>3 month), non-specific low back pain
* 25- 55 years old
* Have a capacity can understand exercise instructions (Montreal Cognitive Assessment > 21)
* Being a computer literate

Exclusion Criteria:

* Root nerve signs
* Cauda equina syndrome
* Fracture in the vertebra
* Tumour
* Have a neurologic disease
* History of spine surgery
* Knowing motor control exercises
* Visual impairment
* Hearing loss

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain Level at Eight Week and Third Month | At baseline, eighth week and third month
  Full Scale Name: Visual Analog Scale
  Pain change will be measured throughout Study and Follow-up with Visual Analog Scale. This scale is a 100 millimeter line drawn horizontally on an A4 sheet of paper. The left end of the line shows "no pain at all", the right end shows "my pain is as bad as it could be", while the remaining part shows the intermediate values. So minimum score was 0, and maximum score was 100. The patient is asked to mark the severity of the pain on the chart. Validity and reliability were made. The minimal clinical significance difference in chronic low back pain was 20 millimeters.
Change from Baseline Disability Score Level at Eight Week and Third Month | At baseline, eighth week and third month
  Full Scale Name: Turkish version of the Oswestry Disability Index (ODI) (2.0)
  The last reliable and validate Turkish Version of Oswestry Disability Index will be used. This version contains 10 multiple-choice questions that question how low back pain affects a person in his or her daily life. Each question has 6 options. As the disability increases, the score of each problem increases. In the worst case you can get 50 points. The last point is the patient's score 100.
Change in Exercise Adherence Level between Eight Week and Third Month | At eighth week and third month
  The Exercise Adherence Rating Scale (EARS), which evaluates exercise compliance, will be administered 2 times to determine change at eight weeks and third month. This scale consists of 3 parts: A, B, C.
  Section A, consists of 6 items not included in the scale scoring.
  Section B consists 6 items, and every item have five point likert scale and describes how to do the recommended home exercise. Minimum point for this section 0, and maximum point is 24. The higher score shown exercise adherece is high.
  Section C is the section that evaluates the reason for the absence of compliance with the recommended home exercise and contains 10 items, every item have five point likert scale. Sections are calculated to result in a possible score between 0 and 40. The higher score shown exercise adherece is high.

SECONDARY OUTCOMES:
Change from Baseline Walking Parameters at Eight Week and Third Month | At baseline, eighth week and third month
  Mean Step Length and Total Walking Distance in Six Minute Walk Test

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03984903/Prot_SAP_000.pdf